CLINICAL TRIAL: NCT03724201
Title: Delirium Severity, Subsyndromal Delirium, and Inflammation-associated Biomarkers in Mechanically Ventilated Patients With Sepsis
Brief Title: Neuronal Damage In Delirium Study
Acronym: NDID
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Kirsten Fiest, PhD, University of Calgary
Other Study IDs: REB18-0409
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Delirium
Keywords: Delirium; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; Neurocognitive Disorders; Mental Disorders; Biomarkers; Pathophysiology
MeSH Terms: conditions — Delirium; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum will be isolated from venous blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate associations between neuronal damage biomarkers (S100 calcium-binding protein beta [S-100β], neuron-specific enolase [NSE], ubiquitin carboxy-terminal hydrolase L1 [UCHL1], and brain-derived neurotropic factor [BDNF]) and delirium severity and subsyndromal delirium in a homogeneous population of mechanically ventilated patients with sepsis.

DETAILED DESCRIPTION:
Due to high levels of inflammation, patients with sepsis are especially at risk of developing delirium, an organic state of confusion that affects over 80% of mechanically ventilated patients during their intensive care stay. A growing body of literature suggests that the severity of delirium symptoms may also have a significant impact on negative outcomes associated with delirium, including mortality, length of hospital stay, duration of mechanical ventilation, and functional and cognitive impairment. Similarly, recent literature suggests that patient outcomes may be worsened by a subthreshold severity level of delirium, known as subsyndromal delirium. Despite the urgent need to understand delirium and subsyndromal delirium etiology for better detection and management strategies, the multifactorial pathophysiology of delirium is still largely unknown. Clinical biomarker studies evaluating levels of S100 calcium-binding protein beta (S-100β), neuron-specific enolase (NSE), ubiquitin carboxy-terminal hydrolase L1 (UCHL1), and brain-derived neurotropic factor (BDNF) have suggested evidence for their role in delirium pathophysiology, but significant associations with delirium severity and subsyndromal delirium have not been reliably established. Evaluating the dose-response relationship of S-100β, NSE, UCHL1, and BDNF with delirium severity and subsyndromal delirium in a homogeneous population of mechanically ventilated patients with sepsis will provide novel insight on the etiological pathway of delirium. The investigators will evaluate effect modification and confounding by inflammation and blood-brain barrier permeability by measuring well-established biomarkers, interleukin-6 (IL-6) and E-selectin, respectively. Understanding the role of neuronal damage in delirium may be a promising avenue to develop better screening practices and neuroprotective management strategies that may reduce long-term cognitive and functional deficits associated with delirium.

ELIGIBILITY:
Inclusion Criteria:

* Located in FMC ICU
* Able to consent or have a surrogate decision-maker able to consent
* Richmond Agitation and Sedation Scale Score ≥ -3
* Glasgow Coma Scale (GCS) score ≥ 9
* Able to communicate with the study team (English language, no hearing impairments)
* Expected to remain in the ICU longer than 24 hours
* Sequential Organ Failure Assessment (SOFA) score ≥2 (indicates sepsis based off of Sepsis 3 Guidelines)
* Invasively mechanically ventilated

Exclusion Criteria:

Neurological injury or neurodegenerative condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients with sepsis will be recruited from the largest adult ICU in Calgary, Alberta Foothills Medical Centre (FMC).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Delirium severity and subsyndromal delirium | Up to five days
  The Confusion Assessment Method for the Intensive Care Unit 7 (CAM-ICU-7) will be completed once per day by a trained research assistant. The CAM-ICU-7 evaluates features and severity of delirium, including 1) acute onset or fluctuating course; 2) inattention; 3) disorganized thinking; and 4) altered level of consciousness. Features 1 and 2, and 3 or 4 must be present to indicate delirium. A non-zero score that does not meet the criteria of delirium indicates subsyndromal delirium. Feature 1 is scored dichotomous (0 or 1), while features 2, 3, and 4 are scored ranging between 0 and 2 (minimum 0, maximum 7). Higher scores indicate more severe delirium or subsyndromal delirium on delirium- or subsyndromal delirium-positive assessments.
Serum concentrations of serum S-100β, NSE, UCHL1, BDNF, E-selectin, and IL-6 | Once on the first day of enrollment
  A serum sample will be collected and processed for batched analysis on the first day of participant enrollment. Serum concentrations of target biomarkers will be quantified using Addressable Laser Bead Immunoassay (ALBIA), a high throughput immunosorbent assay that measures emissions from fluorescently labelled microbeads complexed with antigen-specific capture antibodies to yield a continuous measure of analyte concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten M Fiest, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description — http://cumming.ucalgary.ca/labs/calgary-critical-care-research-network/research/ongoing-projects/ndid-summary